CLINICAL TRIAL: NCT01101256
Title: Determination of Residual Anticoagulatory Effects of Prophylactic or Therapeutic Treatment With Fondaparinux
Brief Title: Determination of Residual Anticoagulatory Effects of Fondaparinux
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Dr. Marc Schindewolf, Division of Vascular Medicine, Department of Internal Medicine, J.W.Goethe University Hospital Frankfurt/Main, Germany
Other Study IDs: 66/09
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Anticoagulant Prophylaxis/Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Citrated blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fondaparinux Prophylaxis group
- Fondaparinux Therapy group

SUMMARY:
The purpose of this study is to determine residual anticoagulatory effects of a prophylactic or therapeutic fondaparinux treatment i.e. prior to surgery/intervention, after pause of therapy etc.

ELIGIBILITY:
Inclusion Criteria:

* Fondaparinux therapy for at least 3 days

Exclusion Criteria:

* Age < 18 years
* Hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with s.c. anticoagulant therapy (fondaparinux)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-09 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
antiXa-levels (peak- and through-levels) | between day 3 and day 14 after start of therapy

SECONDARY OUTCOMES:
thromboembolic or bleeding episodes, HIT | day 14 after start of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schindewolf, MD, Principal Investigator — J.W. Goethe University Hospital Frankfurt/M.
Locations (1):
- J.W. Goethe University Hospital Frankfurt/M., Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Paolucci F, Frasa H, Van Aarle F, Capdevla A, Clavies MC, van Dinther T, Donat F, Hendriks Y, van den Heuvel M, Nadal T, Lagrange F, Necciari J, Perez Y. Two sensitive and rapid chromogenic assays of fondaparinux sodium (Arixtra) in human plasma and other biological matrices. Clin Lab. 2003;49(9-10):451-60. PMID 14572200